CLINICAL TRIAL: NCT03841045
Title: Unraveling a Potential Connection Between Bilirubin Metabolism, Gut Microbiota and Inflammatory Bowel Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, ARIK SEGAL MD, principal investigator, Soroka University Medical Center
Other Study IDs: 0148-15 SOR
Record Dates: First submitted 2018-09-05; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Colitis, Ulcerative; Crohn Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — every enrolled people is asked to give saliva, skin and stool samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ulcerative colitis patient: people that have UC diagnosis can participate in the study. the disease can be at any level and the patients can handle any medications.
- CD patient: people that have CD diagnosis can participate in the study. the disease can be at any label and the patients can handle any medications.
- Health people: control group. no IBD patients can be included. patients with other diseases can be included.

SUMMARY:
Inflammatory Bowel Diseases (IBDs) are a set of recurrent inflammatory conditions that include the colon and small intestine. The two principal conditions include Crohn's disease (CD) and ulcerative colitis (UC). The etiology of which is likely to stem from the interplay of gut microbial imbalances and host. In this study stool cultures, saliva and skin samples will be taken from all participants.

DETAILED DESCRIPTION:
Recent studies have shown that certain CD patients harbor microbial communities that are distinct from those of healthy individuals. These studies suggest a central role of the gut microbial population in CD. The high complexity of the gut microbiome, which is the most densely populated bacterial niche, makes the identification of these bacteria a significant challenge. The bacterial population is comprised from 1013 - 1014 individuals, all belonging roughly to a thousand different species, mostly anaerobic, and most of them (roughly 70% - 80%) are uncultivable.

The goals of this project are to examine a potential link between bilirubin metabolism and IBD, by comparing fecal extracts from healthy humans and IBD patients, and to investigate the underlying mechanism explaining these differences.

ELIGIBILITY:
Inclusion Criteria:

* UC
* CD
* healthy Volunteers

Exclusion Criteria:

• N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: people that have UC, CD diagnosis and healthy can participate in the study. the disease can be at any level and the patients can handle any medications.
  each participant will give fresh stool, saliva and skin samples during the study. only one visit is planned in the study-for sighning ICF and returning samples.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-09-14 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
change of bilirubin metabolism in fecal samples | an average of 1 year after recruitment
  liquid chromatography / mass spectrometric (LCMS) analysis is applied to bilirubin metabolism comparison between IBD patients and healthy humans in fecal extracts
microbial diversity of fecal matter | an average of 1 year after recruitment
  16S rRNA sequencing, is used to compare the microbial diversity between healthy individuals and IBD patients

CONTACTS AND LOCATIONS:
Overall Officials: ARIK SEGAL, MD, Principal Investigator — SOROKA MC
Locations (1):
- soroka MC, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No